CLINICAL TRIAL: NCT06048822
Title: Project Rally: Enhancing Cancer Survivorship With Pickleball
Brief Title: Enhancing Cancer Survivorship With Pickleball
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22455
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer Survivors (Experimental): Participation will last approximately 4-6 months. Participants will be encouraged to attend Pickleball sessions at the YMCA at least twice a week. Each session will last 2 hours, and participants will be encouraged to attend at least one hour. Participants will receive a Fitbit to wear continuously 24/7 over 4-6 months to track steps and activity intensity. Participants will also be asked to wear an electronic device (accelerometer) over their right hip during specific time points throughout the study to better understand how pickleball participation contributes to physical activity levels.
  Interventions: Behavioral: Pickleball
- Family or Friend of Cancer Survivors (Experimental): Participation will last approximately 4-6 months. Participants will be encouraged to attend Pickleball sessions at the YMCA at least twice a week. Each session will last 2 hours, and participants will be encouraged to attend at least one hour. Participants will receive a Fitbit to wear continuously 24/7 over 4-6 months to track steps and activity intensity. Participants will also be asked to wear an electronic device (accelerometer) over their right hip during specific time points throughout the study to better understand how pickleball participation contributes to physical activity levels.
  Interventions: Behavioral: Pickleball

INTERVENTIONS:
Behavioral: Pickleball — Participants will be encouraged to attend ≥2 pickleball sessions per week, with the YMCA offering 5 sessions per week. Sessions will last 2 hours, with participants encouraged to attend ≥1 hour. New players will receive instruction from a YMCA exercise trainer with a USA Pickleball Association Instructor Certification during sessions. At the end of each session, the YMCA trainer will note on attendance sheets whether participants engaged in training/skill development, open play, or both. Participants will be encouraged to engage in 5-10 minutes of structured warm-up exercise (i.e., walking laps around the courts and dynamic and static muscle stretches) prior to playing in each session, and they will be encouraged to perform cool-down stretches after they complete each session.

SUMMARY:
The purpose of the study is to evaluate the feasibility and acceptability of a pickleball program for cancer survivors and their family members or friends. The program is designed to increase physical activity, improve wellness, and allow individuals to work together to learn and practice the sport.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* History of a cancer diagnosis excluding squamous and basal cell skin cancers
* Able to speak and read English
* Able to provide informed consent
* Able to pass a 2023 Physical Activity Readiness Questionnaire+ (PAR-Q+) (with appropriate physician clearance(s), as necessary)
* History of cancer diagnosis will be required for cancer survivor group; friend or family partners can be (but do not need to be) cancer survivors.

Exclusion Criteria:

* Screen failure for exercise safety based on 2023 PAR-Q+
* For cancer survivor group, history of squamous and basal cell skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Recruited - Feasibility | 12 months
  The study will be deemed feasible if ≥ 50% of eligible participants are enrolled
Number of Participants who Complete Baseline Data Collection and Follow up Data Collection - Feasibility | 6 months
  The study will be deemed feasible if ≥ 75% of participants who complete baseline measures also complete follow up measures
Average Pickleball Session Attendance - Feasibility | 6 months
  The study will be deemed feasible if participants attend ≥ 75% of recommended sessions on average.
Participant Evaluation of Feasibility and Acceptability - Acceptability | 6 months
  Participants evaluation of feasibility and acceptability will be assessed with a questionnaire, adapted to fit the intervention. The questionnaire includes both Likert Scale and open-ended questions. An item-by-item basis and as average item score, with scores ≥4 ("agree" to "strongly agree") indicating acceptability. Open-ended responses will be analyzed qualitatively to inform intervention improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Parker, PhD, MPH, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://www.moffitt.org/clinical-trials-and-studies/clinical-trial-22455/